CLINICAL TRIAL: NCT06813248
Title: Effect of Jigsaw Technique on Learning Knowledge About Stroke Patient Care in Nursing Students
Brief Title: Jigsaw Technique and Stroke Patient Care
Status: Recruiting | Type: Observational
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: Burcu Bayrak 2
Record Dates: First submitted 2024-12-20; First posted 2025-02-06 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2024-12

CONDITIONS: Nursing; Education

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the literature, problem-based learning, case discussions and case scenarios, and simulation applications are used in stroke patient care nursing education. However, the use of the jigsaw technique is quite limited. Based on this information, it is anticipated that stroke patient care education provided with the Jigsaw technique can increase nursing students' cooperation and communication skills, allowing them to acquire more effective and comprehensive knowledge in clinical care.

DETAILED DESCRIPTION:
Nursing plays a critical role in protecting the health of individuals and society, preventing diseases and managing health problems. The quality of health services largely depends on the training of qualified nurses. Therefore, effective nursing education is very important for nurses to perform these duties in the best way possible. The effectiveness of the education process directly affects the quality of health services by shaping the knowledge, skills and attitudes of nurses. Innovations and technological advances in the field of medicine have made nursing education a constantly changing and developing field. Traditional education methods have given way to modern, interactive and student-centered approaches. These new approaches in nursing education enable students to gain critical thinking skills; they increase their clinical performance and knowledge adequacy. Many teaching strategies such as simulation applications, problem-based teaching, case discussion, virtual reality, puzzles, concept maps, flipped classrooms, collaborative learning and jigsaw techniques have been incorporated into nursing education. In the jigsaw technique, students form a group and follow a path where each group member learns a part of the subject and shares it with their peers. This means that all students are both learners and teachers in the learning process. Students cooperate and communicate with each other to learn the entire subject, and in this way, the subject is learned completely. The jigsaw technique helps students express their perspectives effectively, actively participate in the learning process, and develop their successes, skills, and positive attitudes. With this method, an active learning environment is created where students support each other and can identify and complete deficiencies. The effective application of this technique significantly increases students' self-confidence, communication skills, problem-solving skills, attitudes towards learning, motivation, sense of responsibility, academic achievements, and retention of information. In the care of stroke patients, nurses' ability to perform a complete neurological assessment, symptom control, and critical thinking skills during the treatment process protect both the physical and psychological well-being of patients, increasing the coordination of the treatment process and patient safety. In addition, effective communication provides support to the family by strengthening not only the harmony within the team but also the harmony of patients and their relatives. Learning information about stroke patient care, developing communication and problem-solving skills, and critical and holistic thinking skills are gained during the nursing education process. Although problem-based learning, case discussions and case scenarios, and simulation applications are used in stroke patient care nursing education in the literature, the use of the jigsaw technique is quite limited. Based on this information, it is anticipated that stroke patient care education provided with the Jigsaw technique can increase the cooperation and communication skills of nursing students and enable them to obtain more effective and comprehensive knowledge in clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Those who were attending class at the time the research data were collected,
* had not received any previous training in stroke patient care,
* agreed to participate in the research

Exclusion Criteria:

* Absenteeism from class

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Nursing students
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
The knowledge level of students on stroke patient care | 15/12/2024-31/01/2025
  As the first outcome of the study, the knowledge level of students on stroke patient care will be measured. A questionnaire consisting of 20 items prepared by the researchers and whose content validity was measured will be used to measure the knowledge level. Each question in the questionnaire will be 5 points and a total of 100 points will be obtained. As the score increases, it will be concluded that the knowledge level is high.
The academic self-efficacy | 15/12/2024-31/01/2025
  As the second outcome of the study, the academic self-efficacy of the students will be measured. For this, the Academic Self-Efficacy Scale for Nursing Students will be used. The scale consists of 14 items and four sub-dimensions in 5-point Likert type. As the score obtained from the scale increases, it is determined that the self-efficacy is high.
The effect of the jigsaw technique on knowledge and academic self-efficacy | 15/12/2024-31/01/2025
  The effect of the jigsaw technique on knowledge and academic self-efficacy. The group learning stroke patient care with the jigsaw method will be compared with the group learning with standard education. The level of knowledge and academic self-efficacy between the two groups will be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Bilecik Seyh Edeabli University, Bilecik, Turkey (Türkiye)